CLINICAL TRIAL: NCT03584763
Title: Frequency of Performing Umbilical Artery Doppler in the Third Trimester in High Risk Pregnancy A Randomized Controlled Trial
Brief Title: Frequency of Performing Umbilical Artery Doppler in the Third Trimester in High Risk Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Hamed Salama, Lecturer of Obstetrics and Gynaecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HRD2010; NCT03562598 (obsolete NCT alias)
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: High Risk Pregnancy

STUDY DESIGN:
Intervention Model Description: Our randomized controlled study was conducted on patients with high risk pregnancies at their third trimester who attended Ain Shams University Maternity Hospital. A total of 292 high risk pregnant women fulfilling the inclusion criteria were selected by random sampling and divided between two groups with 146 patients in each group. Group I underwent Doppler every other week and Group II underwent Doppler once weekly
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding of the patients or staff in this study is not generally feasible. However, the measured outcomes in this study are objective and are unlikely to be biased by lack of blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bi-Weekly Umbilical Artery Doppler (Active Comparator): will undergo Doppler every other week
  Interventions: Diagnostic Test: Umbilical artery Doppler
- Weekly Umbilical Artery Doppler (Experimental): will undergo Doppler every week
  Interventions: Diagnostic Test: Umbilical artery Doppler

INTERVENTIONS:
Diagnostic Test: Umbilical artery Doppler — Umbilical artery Doppler ultrasound will be performed by most expert sonographer in umbilical artery Doppler at the special care unit, using a 3.5MHz transabdominal probe of SAMSUNG MEDISON, SONOACE R5 ultrasound machine, using the standard protocol of the unit for minimizing the interobserver variations.

SUMMARY:
The aim of the current study was to produce a high quality evidence on the best frequency of performing umbilical artery Doppler for high risk pregnant women in the third trimester.

DETAILED DESCRIPTION:
Nowadays, high risk pregnancy forms a significant increasing proportion of any pregnant population, according to some authors up to 50% of all pregnancies would have the label of high risk pregnancies.

At present, it is recommended that high risk pregnancies, thought to be at risk of placental insufficiency should be monitored with Doppler studies of the umbilical artery. Doppler assessment of the placental circulation plays an important role in screening for impaired placentation and its complications of intrauterine growth restriction.

The purpose of umbilical artery Doppler surveillance is to predict fetal academia thereby allowing timely delivery prior to irreversible end-organ damage and intrauterine fetal death.

According to a Cochrane Pregnancy and Childbirth Group's systematic review and meta-analysis, in which Published and unpublished randomised and quasi-randomised trials evaluating the effects of one or more described antenatal fetal surveillance regimens were searched, the optimal frequency of umbilical artery Doppler surveillance is unclear.

Our randomized controlled study was conducted on patients with high risk pregnancies at their third trimester who attended Ain Shams University Maternity Hospital. A total of 292 high risk pregnant women fulfilling the inclusion criteria were selected by random sampling and divided between two groups with 146 patients in each group. Group I underwent Doppler every other week and Group II underwent Doppler once weekly.

ELIGIBILITY:
Inclusion Criteria:

* I-Singleton pregnancy. II-In the third trimester (starting from 28 weeks of gestation till the time of delivery), Gestational age will be determined by the date of the last menstrual period and early ultrasound.

III-Patient considered as high-risk pregnancies will be included in this study.

The following will be considered as high-risk status:

1. Previous obstetric history of preeclampsia or eclampsia, abruptio placenta, intra-uterine growth restriction or still birth.
2. Pre-existing medical disorders like:

   1. Pregestational diabetes (Ang et al., 2006)
   2. Renal diseases (such as nephrotic syndrome, chronic renal failure, renal transplant and hemodialysis) (Divon and Ferber, 2012).
   3. Autoimmune diseases (such as systemic lupus erythromatosis and rheumatoid arthritis) (Divon and Ferber, 2012).
   4. Acquired thrombophilias (such as antiphospholipid syndrome). On the other hand, inherited thrombophilias (such as protein C or S deficiency) are not associated with IUGR (Reeves and Galan, 2012).
   5. Chronic maternal hypoxemia due to pulmonary disease (such as uncontrolled asthma, chronic obstructive pulmonary disease and cystic fibrosis), cardiac disease (such as cyanotic heart disease) or hematologic disorders (such as severe anemia, sickle cell anemia and β-thalassemia) (Baschat et al., 2012).
3. Current preeclampsia or pregnancy-induced hypertension (PIH). PIH is diagnosed in women whose blood pressure reaches 140/90 mm Hg or greater for the first time after midpregnancy, but proteinuria is not identified. Preeclampsia is best described as pregnancy-specific syndrome that can affect virtually every organ system.It is much more than simply gestational hypertension with proteinuria (Cunningham et al, 2010).

IV- Obtaining valid informed consent to participate in the study

Exclusion Criteria:

* I-Patients with congenital anomaly of the fetus. As this will affect fetal outcome with no effect of Doppler changes.

II- Patients with multiple gestations. As they have different growth pattern. III- Patients with unconfirmed Gestational age due to lack of sure reliable date and absent early trimesteric scan. As we cannot diagnose small for gestational age without sure date.

IV- Withdrawal of consent.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 292 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Neonatal admission to r intensive care unit within the first 24 hours | first 24 hours of life
  Neonatal admission to special care and/or intensive care unit within the first 24 hours

SECONDARY OUTCOMES:
Stillbirth | at delivery
  Stillbirth
Neonatal death | 28 days
  Neonatal death
Fetal acidosis | at delivery
  cord blood pH
Apgar score less than seven at five minutes | 5 minutes
  Apgar score less than seven at five minutes
Induction of labour | 24 hours
  Induction of labour
Preterm labour | 37 weeks
  onset of labour before 37 completed week of pregnancy
Gestational age at birth | 28 weeks
  Gestational age at birth
Infant respiratory distress syndrome | 24 hours
  Infant respiratory distress syndrome
Hypoxic ischaemic encephalopathy | 96 hours
  Hypoxic ischaemic encephalopathy
Intraventricular haemorrage | 96 hours
  Intraventricular haemorrage
Necrotizing enterocolitis | 96 hours
  Necrotizing enterocolitis

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf F Nabhan, Professor, Principal Investigator — Faculty of Medicine, Ain Shams University
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
The Investigator will make certain that an appropriate informed consent process is in place to ensure that potential research subjects are fully informed about the nature and objectives of the clinical study, the potential risks and benefits of study participation and their rights as research subjects.
  The Investigator will obtain the written, signed informed consent of each subject prior to performing any study-specific procedures. The Investigator will retain the original signed informed consent form.
  Personal information will not be collected or shared. Unique personal data will be her hospital number.
  Participants files will be maintained in storage for a period of 3 years after completion of the study.

REFERENCES:
- [Result] Alfirevic Z, Roberts D, Martlew V. How strong is the association between maternal thrombophilia and adverse pregnancy outcome? A systematic review. Eur J Obstet Gynecol Reprod Biol. 2002 Feb 10;101(1):6-14. doi: 10.1016/s0301-2115(01)00496-1. PMID 11803092
- [Result] Alfirevic Z, Stampalija T, Gyte GM. Fetal and umbilical Doppler ultrasound in high-risk pregnancies. Cochrane Database Syst Rev. 2013 Nov 12;2013(11):CD007529. doi: 10.1002/14651858.CD007529.pub3. PMID 24222334
- [Derived] Salama MH, Rizk HH, Nawara M. Frequency of third trimester umbilical artery Doppler for improving neonatal outcomes in high-risk pregnancies: a randomized trial. Obstet Gynecol Sci. 2023 May;66(3):161-168. doi: 10.5468/ogs.22130. Epub 2023 Jan 3. PMID 36593702